CLINICAL TRIAL: NCT03117855
Title: A Phase I Clinical Trial of Capecitabine and SIR-Spheres® Y-90-Radioembolization in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Capecitabine and Y-90 Radioembolization in Treating Patients With Advanced Bile Duct Cancer in the Liver That Cannot Be Removed by Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company no longer interested in supporting this trial
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16148; NCI-2016-01098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16148 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-07-27; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bile Duct Adenocarcinoma; Stage III Intrahepatic Cholangiocarcinoma; Stage IVA Intrahepatic Cholangiocarcinoma; Stage IVB Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (capecitabine, yttrium Y-90 radioembolization) (Experimental): Patients undergo yttrium Y 90 resin microspheres radioembolization over 60-90 minutes on day 1. Patients receive capecitabine PO BID on days 1-14.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Radiation: Radioembolization

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radioembolization — Undergo yttrium Y-90 radioembolization
  Other Names: intra-arterial brachytherapy

SUMMARY:
This phase I trial studies the side effects of capecitabine and Y-90 radioembolization in treating patients with bile duct cancer in the liver that has spread to other places in the body and cannot be removed by surgery. Radiation therapy, such as Y-90 radioembolization, injects tiny radioactive Y-90 microspheres into the blood supply next to the liver tumors to kill tumor cells. Capecitabine may make radiation more effective. Giving capecitabine and Y-90 radioembolization may work better in treating patients with bile duct cancer in the liver.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity of capecitabine, to be used in combination with yttrium Y-90 (yttrium 90) (Y-90) radioembolization (RE), in patients with a diagnosis of unresectable intrahepatic cholangiocarcinoma (ICC).

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with Y-90 + capecitabine in patients with ICC.

II. To develop a preliminary assessment of efficacy by evaluating liver-specific progression-free survival (PFS) and overall PFS.

III. To develop a preliminary assessment of efficacy by evaluating response rate according to Response Evaluation Criteria in Solid Tumors (RECIST)/modified RECIST (mRECIST) and the Europeans Association for the Study of the Liver (EASL) imaging criteria.

IV. To develop a preliminary assessment of efficacy by evaluating cancer antigen (CA) 19-9 response and its correlation with imaging markers of tumor response.

V. To develop a preliminary assessment of efficacy by evaluating duration of response in the liver, as measured by the time for target liver lesions to progress according to RECIST/mRECIST beyond size at study enrollment.

VI. To develop a preliminary assessment of efficacy by evaluating rate of conversion to surgical resection for subjects who are surgically unresectable at presentation due to size or location of hepatic lesions (excluding subjects with extrahepatic disease or medically inoperable at presentation).

VII. To develop a preliminary assessment of efficacy by evaluating overall survival.

OUTLINE:

Patients undergo yttrium Y 90 resin microspheres radioembolization over 60-90 minutes on day 1. Patients receive capecitabine orally (PO) twice daily (BID) on days 1-14.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Eastern Cooperative Oncology Group performance status 0-2
* Life expectancy > 3 months
* Intrahepatic cholangiocarcinoma; a histological diagnosis is mandated; a diagnosis of adenocarcinoma with staining pattern consistent with cholangiocarcinoma and with a clinical presentation consistent with cholangiocarcinoma will be acceptable for enrollment as this is a typical intrahepatic cholangiocarcinoma presentation
* Primary tumor deemed unresectable by hepatobiliary surgeon
* Absence of the following:

  * Malignant ascites
  * Extensive carcinomatosis (in the opinion of the investigator)
  * Bulky, diffuse adenopathy (> 5 lymph nodes > 2 cm each)
  * Extensive metastatic disease to the lungs (> 5 tumors > 2 cm each)
* Has completed pre-RE angiogram up to 3 weeks prior to Y-90 therapy

  * Lung shunt fraction =< 20% and anatomy amenable to intra-arterial radiation delivery
  * Extrahepatic vessels deemed at risk for radiation injury were successfully embolized
* Prior systemic chemotherapy must be completed > 2 weeks of radioembolization
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only)
* Platelets (PLT) >= 100,000/mm^3
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Creatinine clearance of > 50 mL/min per 24 hour urine collection of the Cockcroft-Gault formula
* Hemoglobin > 9 g/dL
* Total bilirubin < 2 mg/dL
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and until at least 180 days after administration of any study agent; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Prior selective internal radiation to the liver
* Prior warfarin-based therapies within 7 days of capecitabine treatment
* Actively receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Neuropathy >= grade 2 (moderate neuropathy that limits instrumental activities of daily living)
* History of main or lobar portal vein thrombosis
* History of biliary stent, internal biliary drain, or prior procedure compromising the ampulla of Vater (diagnostic endoscopic retrograde cholangiopancreatography [ERCP] is permissible)
* Known dihydropyrimidine dehydrogenase deficiency
* History of allergic reactions attributed to:

  * Study agent or its metabolites
  * Iodinated contrast media
* Pregnant or breastfeeding (women)
* Concurrent diagnosis of other active malignancies with the exception of ductal carcinoma in situ, cervical carcinoma in situ, and localized non-melanoma skin cancer
* Any clinically significant uncontrolled illness including ongoing active infection
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) defined as any grade 3 or above toxicity assessed by the National Cancer Institute Common Terminology for Adverse Events version 4.0 | Up to day 45
  The toxicities observed at each dose level will be summarized in terms of type, severity, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities. Tabular and graphical summaries will be used to explore the relationship of type and grade toxicity to other clinical parameters such as disease response and the presence of other comorbidities.

SECONDARY OUTCOMES:
Duration of response according to RECIST v1.1, mRECIST, and EASL criteria | Time until tumors progress beyond the values measured at baseline, assessed up to 48 months
  Duration of response will be calculated independently of PFS in order to evaluate the possibility that progression may occur after an initial tumor shrinkage.
Levels of CA 19-9 response | Up to 48 months
  CA 19-9 will be assessed after Y-90 and will be compared to other measures of disease response using Pearson correlation or similar methods.
Liver-specific PFS according to RECIST v1.1, mRECIST, and EASL criteria | Time until tumors progress beyond the values measured at baseline, assessed up to 48 months
  Evaluated using Kaplan-Meier analysis.
Overall survival | Up to 48 months
  Evaluated using Kaplan-Meier analysis.
PFS according to RECIST v1.1, mRECIST, and EASL criteria | Time until tumors progress beyond the values measured at baseline, assessed up to 48 months
  Evaluated using Kaplan-Meier analysis.
Rate of conversion to surgical candidacy | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kessler, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States